CLINICAL TRIAL: NCT01069289
Title: A Phase III, 12-week, Double-blind, Randomised, Parallel-group, Active-controlled, Multinational, Efficacy and Safety Study of Symbicort® Turbuhaler® 160/4.5 μg 2 Inhalations Twice Daily (Bid) Compared to Oxis® Turbuhaler® 4.5 μg 2 Inhalations Twice Daily (Bid) in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Efficacy and Safety Study of Symbicort® Turbuhaler® Versus Oxis® Turbuhaler® in Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: SUMIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D589DC00007
Record Dates: First submitted 2010-02-11; First posted 2010-02-17 (Estimated); Results first posted 2012-10-25 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Symbicort; Oxis; Chronic Obstructive Pulmonary Disease; COPD; Efficacy
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Symbicort Turbuhaler 160/4.5 microgram, 2 inhalations twice daily
  Interventions: Drug: Budesonide/formoterol (Symbicort Turbuhaler)
- 2 (Active Comparator): Oxis Turbuhaler 4.5 microgram, 2 inhalations twice daily
  Interventions: Drug: Formoterol (Oxis Turbuhaler)

INTERVENTIONS:
Drug: Budesonide/formoterol (Symbicort Turbuhaler) — 2x160/4.5 microgram, inhalation, twice daily, 12 weeks
  Other Names: Symbicort Turbuhaler
  Arms: 1
Drug: Formoterol (Oxis Turbuhaler) — 2 X 4.5 microgram, inhalation, twice daily, 12 weeks
  Other Names: Oxis Turbuhaler
  Arms: 2

SUMMARY:
The primary purpose of the study is to investigate if Symbicort is more effective than Oxis in increasing forced expiratory volume in one second (FEV1), measured at the clinics, in patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* A current clinical diagnosis of Chronic Obstructive Pulmonary Disease
* Documented Chronic Obstructive Pulmonary Disease symptoms for more than 2 years
* A smoking history of at least 10 pack years

Exclusion Criteria:

* History and/or current clinical diagnosis of asthma
* History and/or current clinical diagnosis of atopic diseases such as allergic rhinitis

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1293 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Göran Carlsson, MD, Study Chair — AstraZeneca R&D, Lund, Sweden; Yoshinosuke Fukuchi, M.D., PhD, Principal Investigator — Department of Respiratory medicine, Juntendo University
Locations (119):
- India (7):
  - Research Site, Bangalore, Karnataka
  - Research Site, Mysore, Karnataka
  - Research Site, Trivandrum, Kerala
  - Research Site, Indore, Madhya Pradesh
  - Research Site, Nagpur, Maharashtra
  - Research Site, New Delhi, National Capital Territory of Delhi
  - Research Site, Coimbatore, Tamil Nadu
- Japan (62):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Okazaki, Aichi-ken
  - Research Site, Seto, Aichi-ken
  - Research Site, Toyota, Aichi-ken
  - Research Site, Toyota-shi, Aichi-ken
  - Research Site, Akita, Akita
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Yanagawa, Fukuoka
  - Research Site, Gifu, Gifu
  - Research Site, Takayama-shi, Gifu
  - Research Site, Maebashi, Gunma
  - Research Site, Ōta, Gunma
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Obihiro, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Tomakomai, Hokkaido
  - Research Site, Himeji, Hyōgo
  - Research Site, Itami, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Naka-gun, Ibaragi
  - Research Site, Hitachi, Ibaraki
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Sakaidechō, Kagawa-ken
  - Research Site, Kagoshima, Kagoshima-ken
  - Research Site, Fujisawa, Kanagawa
  - Research Site, Kawasaki-shi, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Zama-shi, Kanagawa
  - Research Site, Kochi, Kochi
  - Research Site, Kyoto, Kyoto
  - Research Site, Matsusaka-shi, Mie-ken
  - Research Site, Murata, Miyagi
  - Research Site, Sendai, Miyagi
  - Research Site, Chino-shi, Nagano
  - Research Site, Matsumoto, Nagano
  - Research Site, Isahaya-shi, Nagasaki
  - Research Site, Nagaoka, Niigata
  - Research Site, Saiki-shi, Oita Prefecture
  - Research Site, Yufu-shi, Oita Prefecture
  - Research Site, Kurashiki-shi, Okayama-ken
  - Research Site, Okayama, Okayama-ken
  - Research Site, Urasoe-shi, Okinawa
  - Research Site, Izumi-shi, Osaka
  - Research Site, Kishiwada, Osaka
  - Research Site, Moriguchi, Osaka
  - Research Site, Osaka, Osaka
  - Researche Site, Sakai-shi, Osaka
  - Research Site, Saga, Saga-ken
  - Research Site, Kitakatsushika-gun, Saitama
  - Research Site, Koshigaya-shi, Saitama
  - Research Site, Matsue, Shimane
  - Research Site, Chūō, Tokyo
  - Research Site, Itabashi-ku, Tokyo
  - Research Site, Meguro City, Tokyo
  - Research Site, Minato-ku, Tokyo
  - Research Site, Setagaya City, Tokyo
  - Research Site, Shinagawa-ku, Tokyo
  - Research Site, Suginami-ku, Tokyo
  - Research Site, Sumida-ku, Tokyo
  - Research Site, Wakayama, Wakayama
- Philippines (6):
  - Researche Site, San Fernando City, Pampanga
  - Research Site, Davao City, Philippines
  - Research Site, Iloilo City
  - Research Site, Lipa City, Batangas
  - Research Site, Olongapo City
  - Research Site, Quezon City
- Poland (21):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Chodzież
  - Research Site, Jarosław
  - Research Site, Karpacz
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Loma
  - Research Site, Lublin
  - Research Site, Ostrów Wielkopolski
  - Research Site, Piła
  - Research Site, Poznan
  - Research Site, Ruda Śląska
  - Research Site, Słupca
  - Research Site, Tczew
  - Research Site, Torun
  - Research Site, Turek
  - Research Site, Włoszczowa
  - Research Site, Zabrze
  - Research Site, Zawadzkie
  - Research Site, Żnin
- Russia (7):
  - Research Site, Barnaul, Russia
  - Research Site, Kazan', Russia
  - Research Site, Moscow, Russia
  - Research Site, Saint Petersburg, Russia
  - Research Site, Yekaterinburg, Russia
  - Research Site, Novosibirsk
  - Research Site, Vladikavkaz
- South Korea (3):
  - Research Site, Ansan
  - Research Site, Incheon
  - Research Site, Seoul
- Taiwan (4):
  - Research Site, Chiayi City
  - Research Site, Kaohsiung City
  - Research Site, Keelung
  - Research Site, Taipei
- Ukraine (7):
  - Research Site, Dnipropetrovsk
  - Research Site, Donetsk
  - Research Site, Kyiv
  - Research Site, Poltava
  - Research Site, Uzhhorod
  - Research Site, Vinytsa
  - Research Site, Zaporozye
- Vietnam (2):
  - Research Site, Ho Chi Minh City, Vietnam
  - Research Site, Hanoi

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant entered the study on 28 January 2010, and the last participant completed the study on 30 March 2011. A total of 1,710 participants were enrolled at 163 centres in 9 countries in Asia and Europe, and 1,293 participants who fulfilled the randomisation criteria were randomised.
Pre-assignment Details: The study started with an enrolment visit, Visit 1, 0 to 4 weeks prior to Visit 2, and 1-2 week run-in period before randomization. At Visit 2 participants had to have pre-bronchodilatory forced expiratory volume in one second (FEV1) less than or equal to 50 percent of the predicted normal value.
Groups:
- Symbicort Turbuhaler (Experimental): Symbicort Turbuhaler 160/4.5 microgram (mcg), 2 inhalations twice daily (bid)
- Oxis Turbuhaler (Active Comparator): Oxis Turbuhaler 4.5 microgram (mcg), 2 inhalations twice daily(bid)
Period: Overall Study
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Started | 636 | 657
Completed | 594 | 601
Not Completed | 42 | 56
Not completed — Withdrawal by Subject | 15 | 26
Not completed — Adverse Event | 21 | 28
Not completed — Eligibility criteria not fulfilled | 2 | 0
Not completed — Severe non-compliance to protocol | 3 | 2
Not completed — Due to deteriorating health condition | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator) | Total
Number analyzed (Participants) | 636 | 657 | 1293
Age Continuous [Mean (Full Range); unit: Years] | 64.5 [40 to 89] | 65.6 [40 to 87] | 65.1 [40 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 64 | 143
  Male | 557 | 593 | 1150

OUTCOME MEASURES:

1. Primary Outcome: Pre-dose Forced Expiratory Volume in One Second (FEV1)
Description: The ratio, expressed as percentage, of the geometric mean of available data for Weeks 0, 4, 8 and 12 to the baseline for each treatment group
Time Frame: Before randomization, 0, 4, 8 and 12 weeks after randomization
Population: The analysis set for efficacy was based on the Full Analysis Set (FAS). Available data represent patients who had both baseline and on treatment data which is required to be included in the analysis.
Measure: Geometric Mean (Full Range); unit: percentage of Baseline
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 618 | 635
percentage of Baseline | 104.6 [37.4 to 311.1] | 101.5 [35.1 to 218.5]

2. Secondary Outcome: 1 Hour Post Dose Forced Expiratory Volume in One Second (FEV1)
Description: as for outcome 1
Time Frame: Before randomization, 0, 4, 8 and 12 weeks after randomization
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: percentage of Baseline
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 635 | 657
percentage of Baseline | 113.9 [55.5 to 336.3] | 111.2 [51.3 to 203.3]

3. Secondary Outcome: Pre-dose Forced Vital Capacity (FVC)
Description: as for outcome 1
Time Frame: Before randomization, 0, 4, 8 and 12 weeks after randomization
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: percentage of Baseline
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 618 | 635
percentage of Baseline | 102.2 [57.3 to 313.8] | 100.9 [61.5 to 347.6]

4. Secondary Outcome: 1 Hour Post-dose Forced Vital Capacity (FVC)
Description: as for outcome 1
Time Frame: Before randomization, 0, 4, 8 and 12 weeks after randomization
Population: The analysis set for efficacy was based on the Full Analysis Set (FAS. Available data represent patients who had both baseline and on treatment data which is required to be included in the analysis.
Measure: Geometric Mean (Full Range); unit: percentage of Baseline
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 635 | 657
percentage of Baseline | 110.1 [62.0 to 262.7] | 108.7 [63.5 to 272.7]

5. Secondary Outcome: Percentage of Participants With Exacerbations
Description: A Chronic Obstructive Pulmonary Disease (COPD) exacerbation was defined as worsening in COPD symptoms requiring treatment with either a course of systemic steroid or hospitalisation. The percentage of participants who had experienced COPD exacerbation at the end of the study for each treatment group.
Time Frame: Daily during 12-week randomization treatment
Population: The analysis set for efficacy was based on the Full Analysis Set (FAS).Available data represent patients who had both baseline and on treatment data which is required to be included in the analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 636 | 657
percentage of participants | 11.9 | 16.9

6. Secondary Outcome: Number of Chronic Obstructive Pulmonary Disease (COPD) Exacerbation
Description: A Chronic Obstructive Pulmonary Disease (COPD) exacerbation was defined as worsening in COPD symptoms requiring treatment with either a course of systemic steroid or hospitalisation. Number of COPD exacerbation during 12-week randomization treatment
Time Frame: Daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Number; unit: event
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 636 | 657
event | 93 | 151

7. Secondary Outcome: Morning Peak Expiratory Flow(PEF)
Description: The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period and daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter/minute (L/min)
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 613 | 637
Liter/minute (L/min) | 4.29 (36.58) | -4.78 (30.61)

8. Secondary Outcome: Evening Peak Expiratory Flow (PEF)
Description: The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period and daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter/minute (L/min)
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 612 | 637
Liter/minute (L/min) | 2.55 (36.57) | -5.13 (31.52)

9. Secondary Outcome: Total Number of Day With Exacerbation
Description: Total number of days with COPD exacerbation for each treatment group
Time Frame: Daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Number; unit: days
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 636 | 657
days | 653 | 1098

10. Secondary Outcome: Morning Forced Expiratory Volume in One Second (FEV1)
Description: The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period and daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 613 | 637
Liter (L) | 0.0244 (0.2136) | -0.0312 (0.1712)

11. Secondary Outcome: Evening Forced Expiratory Volume in One Second (FEV1)
Description: The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period and daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 612 | 637
Liter (L) | 0.0176 (0.2268) | -0.0324 (0.1724)

12. Secondary Outcome: Night-time Awakening Due to Chronic Obstructive Pulmonary Disease (COPD) Symptoms
Description: Scored 0 to 1 (0 = no awakening and 1 = awakening). The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period and daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Nights with symptoms
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 628 | 647
Nights with symptoms | -0.20 (0.67) | -0.15 (0.66)

13. Secondary Outcome: Breathlessness Due to Chronic Obstructive Pulmonary Disease (COPD) Symptoms
Description: There are 5 alternatives (scored 0 to 4, with 4 being the most severe condition). The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period and daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 628 | 647
units on a scale | -0.34 (0.66) | -0.23 (0.65)

14. Secondary Outcome: Cough Due to Chronic Obstructive Pulmonary Disease (COPD) Symptoms
Description: as for outcome 13
Time Frame: Daily during run-in period and daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 628 | 647
units on a scale | -0.24 (0.70) | -0.24 (0.68)

15. Secondary Outcome: Total Chronic Obstructive Pulmonary Disease (COPD) Symptom Score
Description: The Total COPD Symptom score is the sum of the measures night-time awakening, breathlessness and cough, ranges from 0 to 12 with 12 being the most severe. The change from Run-in period average to Treatment period average for each treatment group.
Time Frame: Daily during run-in period and daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 628 | 647
units on a scale | -0.78 (1.62) | -0.61 (1.56)

16. Secondary Outcome: Use of Rescue Medication
Description: The change from Run-in period average to Treatment period average for each treatment group.
Time Frame: Daily during run-in period and daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: inhalations/day
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 628 | 647
inhalations/day | -0.51 (1.51) | -0.26 (1.49)

17. Secondary Outcome: St George's Respiratory Questionnaire (SGRQ) Total Score
Description: The change from Run-in period average to Treatment period average for each treatment group. The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
Time Frame: Daily during run-in period and daily during 12-week randomization treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Number analyzed (Participants) | 621 | 634
units on a scale | -4.37 (14.544) | -2.90 (13.783)

ADVERSE EVENTS:
Arm/Group | Symbicort Turbuhaler (Experimental) | Oxis Turbuhaler (Active Comparator)
Serious Adverse Events (participants affected / at risk) | 43/636 | 45/657
Other Adverse Events (participants affected / at risk) | 61/636 | 66/657
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort Turbuhaler (Experimental) (N=636) | Oxis Turbuhaler (Active Comparator) (N=657)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 24 | 28
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1 | 2
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 1
INFECTIVE EXACERBATION OF CHRONIC OBSTRUCTIVE AIRWAYS DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 3
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 3 | 1
APPENDICITIS (Infections and infestations) | 2 | 0
PNEUMONIA BACTERIAL (Infections and infestations) | 1 | 1
BRONCHITIS (Infections and infestations) | 0 | 1
BRONCHOPNEUMONIA (Infections and infestations) | 1 | 0
POSTOPERATIVE ABSCESS (Infections and infestations) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 1
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 0 | 1
DIVERTICULUM INTESTINAL HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 1
ILEUS (Gastrointestinal disorders) | 1 | 0
PANCREATIC MASS (Gastrointestinal disorders) | 0 | 1
PERITONITIS (Gastrointestinal disorders) | 1 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
METASTASES TO LUNG (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 1 | 0
CARDIOVASCULAR INSUFFICIENCY (Cardiac disorders) | 1 | 0
CORONARY ARTERY INSUFFICIENCY (Cardiac disorders) | 0 | 1
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1
BRAIN STEM STROKE (Nervous system disorders) | 1 | 0
HYPOXIC-ISCHAEMIC ENCEPHALOPATHY (Nervous system disorders) | 1 | 0
ISCHAEMIC STROKE (Nervous system disorders) | 0 | 1
AMAUROSIS FUGAX (Eye disorders) | 1 | 0
CATARACT (Eye disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0
DEATH (General disorders) | 1 | 0
AORTIC ANEURYSM RUPTURE (Vascular disorders) | 0 | 1
COMPUTERISED TOMOGRAM THORAX ABNORMAL (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort Turbuhaler (Experimental) (N=636) | Oxis Turbuhaler (Active Comparator) (N=657)
Nasopharyngitis (Infections and infestations) | 35 | 32
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 29 | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other